CLINICAL TRIAL: NCT01830517
Title: Comparison of the Effects of Amlodipine and Losartan on Blood Pressure and Diurnal Variation in Hypertensive Stroke Patients
Brief Title: Diurnal Variation in Hypertensive Stroke Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-AMO-401
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension; Stroke
MeSH Terms: conditions — Hypertension; Stroke | interventions — amlodipine-losartan drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- amlodipine camsylate (Experimental): amlodipine camsylate 5mg
  Interventions: Drug: Amlodipine, Losartan
- losartan potassium (Active Comparator): losartan potassium 50mg
  Interventions: Drug: Amlodipine, Losartan

INTERVENTIONS:
Drug: Amlodipine, Losartan

SUMMARY:
This study was conducted to evaluate and compare the effectiveness of Amodipin® (amlodipine camsylate) with that of Cozaar® (losartan potassium) in hypertensive patients with an acute ischemic stroke by measuring their 24-hour ambulatory BP (ABP).

ELIGIBILITY:
Inclusion Criteria:

1. aged 35 to 85 years
2. hypertensive patients who had an ischemic stroke

Exclusion Criteria:

1. patients aged below 35 years or above 86 years;
2. patients who had a hemorrhagic stroke;
3. patients whose systolic BP (SBP) was over 220 mmHg or whose diastolic BP (DBP) was above 120 mmHg during an acute phase, or whose SBP was over 180 mmHg or whose DBP was over 110 mmHg one week after their hospital visit;
4. patients with secondary hypertension related to renovascular, endocrinologic, or pregnant conditions
5. patients who went to bed in the middle of the day or very late at night; (6) patients who were using intravenous antico-agulants or thrombolytics;

(7) patients with a severe stroke (NIH stroke scale > 20); (8) patients who could not give their consent to investigators; (9) patients with severely impaired liver function (AST or ALT ≥ 100); (10) patients with severely impaired renal function (serum creatinine ≥ 2.0 mg/dL); (11) patients with cancer; (12) patients who were pregnant or lactating; (13) patients with other grave diseases such as hypertensive encephalopathy, aortic dissection, acute myocardial infarction, or severe congestive heart failure; and (14) patients who were allergic to the test or control drugs

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory mean SBP | baseline and 8weeks

SECONDARY OUTCOMES:
24H mean DBP, 24H mean SBP/DBP Variability,clinic SBP/DBP, awake, sleep, morning, evening, and prewake BPs, the morning surge, and the nocturnal dipping | baseline and 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyunwoo Nam, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Boramae Medical Center, Boramae-ro 5-gil 20, Dongjak-gu, Seoul, South Korea

REFERENCES:
- [Derived] Kwon HM, Shin JW, Lim JS, Hong YH, Lee YS, Nam H. Comparison of the effects of amlodipine and losartan on blood pressure and diurnal variation in hypertensive stroke patients: a prospective, randomized, double-blind, comparative parallel study. Clin Ther. 2013 Dec;35(12):1975-82. doi: 10.1016/j.clinthera.2013.10.013. Epub 2013 Dec 2. PMID 24296324